CLINICAL TRIAL: NCT01830803
Title: Reliability of howRU and howRwe Questionnaires
Status: Completed | Type: Observational
Sponsor: Medical Research Foundation, The Netherlands (Other)
Responsible Party: Principal Investigator, Henk Bilo, MD, MD PhD, Medical Research Foundation, The Netherlands
Other Study IDs: HowRU/we/1
Record Dates: First submitted 2013-04-05; First posted 2013-04-12 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Quality of Life
Keywords: howRU; howRwe; reliability; quality of life; quality of care; patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HowRU/HowRwe: All participants will fill out the HowRwe and HowRU questionnaires. Although this questionnaire may be considered an intervention, it is not the goal of this study to investigate the questionnaires as an intervention but to investigate whether they are reliable questionnaires.

SUMMARY:
Quality of life and patient satisfaction are two important concepts in health care, especially in chronic diseases. Currently, there are several instruments available to determine this, but many are not easily applicable in daily practice because of their length and the consequential effort they require from both patients and caregivers.

In the UK, Benson et al. recently developed two short generic patient questionnaires on quality of life and patient satisfaction: the howRu and howRwe questionnaires. Both questionnaires contain four items.

The howRU questionnaire has already been validated and seems highly applicable to be used in large patient groups. The howRwe questionnaire has not been validated yet. The reliability of both questionnaires has not been assessed either. The procedure as suggested by Kocks et al. provides us with the opportunity to perform a reliability procedure on patient level.

The purpose of this study is to assess the reliability of the howRU and the howRwe questionnaires on patient level in the Dutch population.

DETAILED DESCRIPTION:
Prior to the start of this study, the howRU and howRwe questionnaires have been translated into Dutch by the MAPI-institute.

All possible eligible patients who are visiting the general practice between February 2013 and April 2013 are asked to complete the howRU questionnaire prior to consultation and the howRwe questionnaire directly after consultation. The scores are not shown to the health care provider who will also complete both questionnaires after consultation as he/she thought the patient should have completed the questionnaires.

An investigator will then select patients based on the scores on the howRU and howRwe questionnaires and their diseases. We will aim to include at least 90 patients: a minimum of 30 patients with diabetes, 30 COPD patients and 30 persons without these diseases. For each patient category, a maximum of 15 patients with a maximum score (defined as 10-12) will be included. All other patients need to have lower scores. As this study aims to assess the reliability of the questionnaires, it is not necessary to select the study participants at random.

The selected patients will be asked to participate in our study. Participating patients will be asked to fill in other questionnaires (EQ-5D and Europep) and the investigator will hold semi-structured interviews, preferably on the day of consultation. Patients are asked to comment on each separate concept of the questionnaires. They are asked what thoughts they had during the completion of the individual questions, and are asked to give examples of these.

The participants' opinions about the questionnaires will also be asked. All interviews will be recorded and fully transcribed. All references to scores on individual items of the questionnaire (in number or words) will be covered with black bars to blind these results. These elaboration will be sent to a reviewing panel consisting of 45 clinicians and 45 patients. They will be instructed to complete the howRU and howRwe questionnaires of a patient, the way they thought the patient should have rated the questionnaires based on the interview, gender and age. Each interview has to be reviewed and scored by five separate clinicians and five patients for both howRU and howRwe.

Each set of interviews, that will be sent out for review, will contain 10 randomly assigned interviews, including information on the patients' gender and age. The order in which interviews will be in the package will be randomised to prevent fatigue of the reviewers and learning effects in the interviews performed later in sequence. Additionally, all interviews will be sent to a panel of patients. These patients will be selected by an investigator.

For statistical analysis SPSS will be used. The data will be manually entered twice to check for errors. The agreement between patient score, treating physician/nurse practitioner and reviewing panel will be presented in Bland & Altman plots for both the howRU and howRwe questionnaires. To assess normality Q-Q plot will be used.

The concordance between patient scores, treating physician/practice nurse scores, and the mean of the scores of the reviewing clinicians and patients will be studied by Lin's concordance correlation (CCC), an extended intraclass correlation (ICC). Additionally, the scores of the five reviewing clinicians will be compared to the scores of the patient panel, also using the ICC.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Visiting the general practice in the period of February/March to May 2013

Exclusion Criteria:

* Illiteracy
* Insufficient understanding of the Dutch language
* Mental retardation
* Visual impairments, such that the questionnaires can not be read

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients visiting a general practice will be asked to participate. We will select patients based on their scores on the howRU and howRwe questionnaires. We will aim to include at least 90 patients: a minimum of 30 patients with diabetes, 30 COPD patients and 30 persons without these diseases.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2013-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Reliability HowRU and HowRwe | Average 12 weeks
  This primary outcome measure concerns the scores on the howRU and howRwe questionnaires as filled out by the patients and the reviewing panel.

SECONDARY OUTCOMES:
HowRU and HowRwe physician scores | 1 day
  The agreement and concordance between patient scores and treating physician/nurse practioner scores on both the howRU and the howRwe questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Jojanneke Rutgers, Bsc, Principal Investigator — Unaffiliated/RUG?; Marco Blanker, MD, PhD, Study Director — University Medical Center of Groningen, department of general practice; Hans van Hateren, MD, PhD, Study Director — Diabetes Center Isala Clinics, Zwolle, the Netherlands
Locations (1):
- General Practice Blanker en Thiele, Zwolle, Overijssel, Netherlands

REFERENCES:
- [Background] Benson T, Sizmur S, Whatling J, Arikan S, McDonald D, Ingram D. Evaluation of a new short generic measure of health status: howRu. Inform Prim Care. 2010;18(2):89-101. doi: 10.14236/jhi.v18i2.758. PMID 21078231
- [Background] Kocks JW, Kerstjens HA, Snijders SL, de Vos B, Biermann JJ, van Hengel P, Strijbos JH, Bosveld HE, van der Molen T. Health status in routine clinical practice: validity of the clinical COPD questionnaire at the individual patient level. Health Qual Life Outcomes. 2010 Nov 16;8:135. doi: 10.1186/1477-7525-8-135. PMID 21080960
- [Derived] Hendriks SH, Rutgers J, van Dijk PR, Groenier KH, Bilo HJ, Kleefstra N, Kocks JW, van Hateren KJ, Blanker MH. Validation of the howRu and howRwe questionnaires at the individual patient level. BMC Health Serv Res. 2015 Oct 2;15:447. doi: 10.1186/s12913-015-1093-8. PMID 26431695